CLINICAL TRIAL: NCT00670930
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled, Parallel-group Trial to Explore the Effects of 78 Weeks Omalizumab Treatment Given as Add on Therapy on Markers of Airway Inflammation and Remodeling in Patients With Moderate to Severe Persistent Allergic Asthma Receiving Inhaled Corticosteroids and Long Acting Beta-agonists
Brief Title: Efficacy of Omalizumab in Adults (18-60 Years of Age) With Moderate-Severe, Persistent Allergic Asthma, Despite Receiving Inhaled Corticosteroids and Long Acting Beta-agonists
Acronym: eXplore
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIGE025A2432; 2007-004653-29 (EudraCT Number)
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-11

CONDITIONS: Allergic Asthma
Keywords: Asthma, adults, anti-immunoglobulin E ( IgE), omalizumab, airway inflammation, airway remodeling, allergy
MeSH Terms: conditions — Asthma; Epilepsy, Idiopathic Generalized; Airway Remodeling; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- omalizumab (Active Comparator): Omalizumab was supplied as lyophilized, sterile powder in a single use, 5 ml vial that was designed to deliver 150 mg of omalizumab for subcutaneous (SQ) administration upon reconstitution with 1.4 ml sterile water for injection. The dose administered was individualized for each patient based on the patient's body weight and total serum Immunoglobulin E (IgE) level at Visit 1 and the number of injections and injection volume was determined using protocol-specified dosing tables. Omalizumab 75 to 375 mg was administered SQ every 2 or 4 weeks depending on the dose for the 78 weeks duration of double-blinded treatment.
  Interventions: Drug: omalizumab at a dose of 0.016mg/kg/IU/mL
- Placebo (Placebo Comparator): Omalizumab matching placebo was supplied as lyophilized, sterile powder in a single-use, 5 ml vial that was designed to deliver omalizumab matching placebo for subcutaneous (SQ) administration upon reconstitution with 1.4 ml sterile water for injection. The number of injections and injection volume was individualized for each patient based on the patient's body weight and total serum Immunoglobulin E (IgE) level at Visit 1 and was determined using protocol-specified dosing tables. Placebo was administered SQ every 2 or 4 weeks for the 78 weeks duration of double-blinded treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: omalizumab at a dose of 0.016mg/kg/IU/mL
  Arms: omalizumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of omalizumab on the number of tissue eosinophils and other markers of airway inflammation and remodeling, including thickness of the lamina reticularis, in moderate to severe asthmatics with persistent symptoms and evidence of airway inflammation despite treatment with inhaled corticosteroids and long acting beta-agonists. This study will also investigate the correlation between systemic and pulmonary inflammation, and the correlation between clinical outcomes and changes within the tissue, to assist in the future identification of patients with tissue eosinophilia and their response to treatment, without the need for invasive bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-75 years of age with moderate to severe persistent allergic asthma receiving a high dose inhaled corticosteroid (≥800µg per day BDP or equivalent) and a regular long acting beta-agonist for at least 3 months prior to screening
* With a body weight between 20 and 150kg and a serum total IgE level of 30 to 700 IU/mL
* With ≥2% eosinophilia in induced sputum at screening
* With post-bronchodilator forced expiratory volume in 1 second (FEV1) ≥60% predicted
* With a positive skin prick test (diameter of wheal ≥ 3 mm) or RAST test to at least one perennial aero-allergen (eg. dust mite, cat/dog dander, cockroaches), documented within the past 2 years or demonstrated at Visit 1, to which the patient will be exposed on a regular basis (most days) for the duration of the study.

Exclusion Criteria:

* Patients who've had an asthma exacerbation during the 4 weeks prior to randomization
* Current smokers, stopped smoking within the last 12 months or have a smoking history of >10 pack years
* History of severe allergy to food or drugs
* Previous treatment with omalizumab
* Any patient considered to be unsuitable to bronchoscopy, according to the judgment of the investigator

Other protocol-defined inclusion/exclusion criteria applied.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (5):
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Galveston, Texas
- Canada (3):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Novartis Investigative Site, Montpellier, France
- Novartis Investigative Site, Mainz, Germany, Germany
- Novartis Investigative Site, Leiden 2333 ZA, Netherlands, Netherlands
- Novartis Investigative Site, Lund, Sweden
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow - Scotland
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton

REFERENCES:
- See also: patient recruitment website — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=664

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 23 ("Started" indicates Randomized and Safety populaiton) | 13
Intent to Treat (ITT) Population | 23 | 12
Completed | 22 | 12
Not Completed | 1 | 1
Not completed — Adminstrative Problem | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 23 | 12 | 35
Age Continuous [Mean (Standard Deviation); unit: Years] — Demographics analysis based on Intent to treat population.
  Years | 43.7 (9.66) | 41.8 (10.43) | 43.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Subepithelial Eosinophils at the End of Week 78 (End of Treatment)
Description: The primary variable of change from baseline in total epithelia eosinophils at end of Week 78 was analyzed on sub-population such as responders and non-responders. Responders are defined as all patients having a Global Evaluation of Treatment Effectiveness (GETE) outcome of excellent or good where as non-responders are with GETE outcome of poor, moderate or worsening. GETE categories are excellent, good, moderate, poor, worsening, and missing as determined by the investigator.
Time Frame: Baseline, at end of week 78
Population: Intent-to-treat (ITT) population: The ITT population consisted of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization. Patients with both baseline and af end of week 78 data in each category have been reported.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 17 | 11
cells/mm^2
  Responder (n= 9, 3) | -5.807 (13.921) | -5.890 (9.128)
  Non-responder (n = 8, 8) | 1.555 (11.065) | -5.626 (15.816)

2. Secondary Outcome: Change From Baseline in Sub-epithelial Cell Count of Mast Cells Following 78 Weeks Treatment, as Assessed Biopsy Samples
Description: The variable of change from baseline in Sub-epithelial cell count of mast cells at end of Week 78 was analyzed on sub-population such as responders and non-responders. Responders are defined as all patients having a Global Evaluation of Treatment Effectiveness (GETE) outcome of excellent or good where as non-responders are with GETE outcome of poor, moderate or worsening. GETE categories are excellent, good, moderate, poor, worsening, and missing as determined by the investigator.
Time Frame: Baseline, at end of week 78
Population: Intent-to-treat (ITT) population: The ITT population consisted of all randomized patients. Patients with both baseline and end of treatment (at the end of week 78) data were only included for the analysis under each category.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 17 | 11
cells/mm^2
  Responder (n= 9, 3) | -1.392 (13.123) | 5.840 (19.809)
  Non-responder (n= 8, 8) | 10.140 (10.266) | 1.114 (18.397)

3. Secondary Outcome: Change From Baseline in Sub-epithelial CD4+ T-lymphocytes Following 78 Weeks Treatment, as Assessed Biopsy Samples
Description: The variable of change from baseline in Sub-epithelial CD4+ T-lymphocytes at end of Week 78 was analyzed on sub-population such as responders and non-responders. Responders are defined as all patients having a Global Evaluation of Treatment Effectiveness (GETE) outcome of excellent or good where as non-responders are with GETE outcome of poor, moderate or worsening. GETE categories are excellent, good, moderate, poor, worsening, and missing as determined by the investigator.
Time Frame: Baseline, at end of week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 17 | 11
cells/mm^2
  Responder (n= 9, 3) | -5.820 (12.490) | -2.693 (8.117)
  Non-responder (n= 8, 8) | -4.719 (11.021) | -7.320 (13.950)

4. Secondary Outcome: Change From Baseline in Thickness of the Lamina Reticularis Following 78 Weeks Treatment, as Assessed Biopsy Samples
Description: The variable of change from baseline in thickness of the lamina reticularis at end of Week 78 was analyzed on sub-population such as responders and non-responders. Responders are defined as all patients having a Global Evaluation of Treatment Effectiveness (GETE) outcome of excellent or good where as non-responders are with GETE outcome of poor, moderate or worsening. GETE categories are excellent, good, moderate, poor, worsening, and missing as determined by the investigator.
Time Frame: Baseline, at end of week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometer(µm)
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 16 | 11
micrometer(µm)
  Responder (n= 8, 3) | -1.300 (2.926) | -1.603 (0.258)
  Non-responder (n= 8, 8) | 0.098 (2.276) | -0.659 (2.288)

5. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death as an Assessment of Safety and Tolerability of 78 Weeks Therapy
Time Frame: 78 weeks
Population: The safety population consisted of all patients in the intent to treat (ITT) population that received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 23 | 13
Participants
  At least one adverse event | 19 | 12
  At least one serious adverse event | 1 | 0
  Death | 0 | 0

ADVERSE EVENTS:
Groups:
- Omalizumab: Omalizumab
- Placebo: Placebo
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/13
Other Adverse Events (participants affected / at risk) | 16/23 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=23) | Placebo (N=13)
Biliary colic (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=23) | Placebo (N=13)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Photopsia (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Injection site erythema (General disorders) | 2 | 0
Injection site rash (General disorders) | 0 | 1
Injection site swelling (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Alveolar osteitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2
Pneumonia (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 2 | 3
Tooth abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.